CLINICAL TRIAL: NCT05111158
Title: Multifocal Electro Retinogram Study of Hydroxy Chloroquine Retinopathy in Lupus Nephritis Patients: A Randomized Controlled Clinical Trial."
Brief Title: MFERG Study of HCQ Retinopathy in Lupus Nephritis Patients: A Randomized Controlled Clinical Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Salah, Doctor, Minia University
Other Study IDs: MFERG in lupus nephritis
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: mfERG in Lupus Nephritis
Keywords: mfERG; HCQ Retinopathy; Lupus nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 50 eyes of 25 SLE patients with renal affection (Lupus nephritis).: mfERG
  Interventions: Diagnostic Test: mfERG
- 50 eyes of 25 SLE patients without renal affection: mfERG
  Interventions: Diagnostic Test: mfERG

INTERVENTIONS:
Diagnostic Test: mfERG — mfERG was performed by RETI Scan (Roland consulting company) and software 6.16.3.10 according to the protocol of the International Society for Clinical Electrophysiology of Vision (ISCEV)

SUMMARY:
The aim of the study to assess the multifocal ERG (mfERG) changes in SLE patients treated with chloroquine in renal patients with comparison to SLE patients without kidney affection.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune inflammatory

disease that involves different organs and systems. The heterogeneous nature of

the disease represents a great challenge in its diagnosis and management.1 Studies

reported that the percentage of SLE patients demonstrating ocular manifestations

can reach up to 30%.2

The pathogenesis of the ocular involvement is still unclear, but immune

complex vasculopathy and inflammatory mediators might be implicated. The most

common ocular manifestation in SLE was found to be kerato-conjunctivitis

sicca(KCS) followed by retinopathy, where is the most severe manifestation was

the optic nerve involvement, which might end up with irreversible blindness while

anterior uveitis is a rare manifestation in SLE.3

Retinal involvement can vary from subclinical vascular changes to vaso-

occlusive vision-threatening retinopathy. Lupus retinopathy is secondary to IgG

complex-mediated micro-angiopathy that leads to small vessels infarcts. Currently,

there is no agreement on existing biomarkers to identify SLE patients who have

subclinical retinal involvement, or to identify whether micro-vascular changes in

the retina are attributable to SLE.4 Lupus retinopathy is usually associated with

high disease activity especially nephritis and cerebritis. 5

On the other side, hydroxychloroquine,(HCQ) a cornerstone in lupus treatment, rarely causes ocular toxicity at doses of less than 6.5 mg/kg per day. Moreover, HCQ is found to be associated with retinopathy after a prolonged time of treatment (>5 years). 6 HCQ bind to melanin pigments in the retinal pigment epithelium (RPE). This binding may serve to concentrate the agents in the cell and contribute to their long-term effects. The classic pattern of retinal toxicity of HCQ is RPE depigmentation with foveal sparing, known as bull's-eye maculopathy. Although visual acuity in these patients seems intact, patients complain from paracentral scotomas associated with reading difficulties. Besides, reduced color perception can be seen as retinopathy symptoms. That is why it is important to evaluate the eyes before starting therapy and during follow-up visits. 7 To diagnose HCQ-induced retinopathy, various methods have been recommended, including: Spectral Domain Optical Coherence Tomography (SD-OCT), automated perimetry test, multifocal electroretinogram (mfERG), But it is controversial as to which of these methods is the Gold Standard early detection of HCQ-induced retinopathy. So it's important to find a tool that can help us diagnose early. 8 mfERG is highly sensitive among the mentioned tests and because it is an objective test, it is less dependent on the patient's response and cooperation .The mfERG objectively evaluates the electroretinographic response of the macular region, and in HCQ retinopathy, this response is reduced in the paracentral region

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old. 2. Emmetropic patients with normal fundus. 3. Patients with SLE diagnosed by a rheumatologist with no ocular involvement upon clinical examination.

Exclusion Criteria:

- 1. Patients with history of intraocular surgery as cataract surgery ,retinal detachment surgery, anti-glucoma surgery.

2. Patients with significant media opacity as corneal opacity, cataract. 3. Patients with ocular diseases as glaucoma, uveitis. 4. Patients with systemic diseases as diabetes mellitus, hypertension.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Residents of Minia Governorate diagnosed with SLE with renal affection and without renal affection.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of mfERG parameters | 3 months
  Analysis of N1, P1, N2 in five concentric areas of the macula between the two groups.
Analysis of values of R1 or R2 amplitude or Ring Ratio | 3 months
  Abnormal values of R1 or R2 amplitude or Ring Ratio (R1 / R2, R1 / R3, R1 / R4, R1 / R5) in each of the patient's eyes as abnormal mfERG.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Salah, MD, Principal Investigator — Minia University Hospital
Locations (1):
- Minia University Hospital, Minya, Egypt